CLINICAL TRIAL: NCT02649972
Title: Phase II Trial of Single-agent Cobimetinib for Adults With Histiocytic Disorders
Brief Title: Single-agent Cobimetinib for Adults With Histiocytic Disorders
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-216
Record Dates: First submitted 2016-01-06; First posted 2016-01-08 (Estimated); Results first posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2022-12

CONDITIONS: Histiocytic Disorders
Keywords: Cobimetinib; 15-216
MeSH Terms: interventions — cobimetinib

ARMS (1):
- Cobimetinib (Experimental): This is an open-label, multicenter, phase II study exploring the efficacy and safety of single-agent Cobimetinib in patients with histiocytic disorders whose tumors are 1) BRAFV600 wildtype or 2) BRAFV600E mutant and are intolerant to, or unable to access, BRAF inhibitors. Visits during the treatment period are to be completed on Day 1, Day 15 (this visit can be by telephone), Day 29, and every 28 days thereafter. For patients treated on the study for six months, at the discretion of the Principal Investigator, visits can be spaced out to every 56 days (every 2 cycles instead of every cycle). After 24 cycles of treatment, if imaging demonstrates sustained stability in the opinion of the principal investigator, tumor assessments can be performed ever 1 year.
  Interventions: Drug: Cobimetinib

INTERVENTIONS:
Drug: Cobimetinib — Cobimetinib will be administered at a dose of 60mg daily for 21 days on, then 7 days off, in a 28 day treatment cycle. Patients will have the option to discontinue treatment after 12 cycles and will be monitored for disease relapse for an additional 12 months. In the event that disease relapse occurs within the 12 month monitoring period, patients will restart treatment and continue on study. Upon restarting, the assessment schedule will restart at rechallenge cycle 1(RC-1) and all assessments will occur at the frequency and intervals. Cycle 1 Day 15 visits will not be required for patients that restart treatment after relapse. Participants will re-sign consent upon rechallenging.

SUMMARY:
The purpose of this study is to find out what effects, good or bad, Cobimetinib has in patients with histiocytosis. Cobimetinib is an investigational oral medication that blocks MEK1.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed histiocytic disorder or histologic findings compatible with a histiocytic disorder in the context of confirmatory radiologic findings confirmed by the enrolling institution.
* One of the following:

  * Documentation of BRAF V600E mutation and inability to access of BRAF inhibitor or prior treatment with a BRAF inhibitor discontinued due intolerable side effects or toxicity prior to progression, -OR-
  * Documentation of wild-type BRAF V600 mutational status
  * Patients with BRAF-mutated ECD/LCH who have had disease progression on BRAF inhibitor therapy would be eligible but would require tissue biopsy (or available tissue) for genotyping before participating.
* Measurable disease according to PET Response Criteria, confirmed by the MSK investigator radiologist, with the exception of patients with cutaneous disease that can be measured and followed by RECIST criteria
* Histiocytic disorder must be (a) multi-system disease or (b) disease that is recurrent or refractory to standard therapies, or (c) single-system disease with that is unlikely to benefit from conventional and less toxic therapies, based on the best available evidence (for example, CNS or cardiac infiltration, retroperitoneal fibrosis, prior chemotherapy, or other medical history or co-morbidities, etc)
* Life expectancy > 12 weeks
* Age ≥ 16 years
* ECOG performance status ≤ 3 (May be converted from Karnofsky Performance Status)
* Adequate bone marrow function as indicated by the following:

  * ANC > 1000/uL
  * Platelets ≥ 50,000/uL
  * Hemoglobin ≥ 8.5 g/dL.
* Patients with cytopenias below these thresholds deemed to be the result of disease will be considered eligible.
* Adequate renal function, as indicated by:

  * creatinine ≤ 1.5 the upper limit of normal (ULN) -OR-
  * Estimated creatinine clearance of > 50 ml/min
* As for #7, patients with renal dysfunction deemed to be the result of disease will be considered eligible.
* Adequate liver function, as defined by bilirubin ≤ 1.5 ULN
* AND AST/ALT < 3 ULN
* Ability to swallow pills
* Negative serum pregnancy test within 7 days prior to commencement of dosing in premenopausal women. Women of non-childbearing potential may be included without serum pregnancy test if they are either surgically sterile or have been postmenopausal for ≥ 1 year.
* Fertile men and women must use an effective method of contraception during treatment and for at least 6 months after completion of treatment as directed by their physician. Effective methods of contraception are defined as those which result in a low failure rate (i.e., less than 1% per year) when used consistently and correctly (for example implants, injectables, combined oral contraception or intra-uterine devices). At the discretion of the Investigator, acceptable methods of contraception may include total abstinence in cases where the lifestyle of the patient ensures compliance. (Periodic abstinence [e.g., calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception.)
* Patients must be willing to consent for protocol #12-245 for IMPACT testing (for MSK patients ONLY).

Exclusion Criteria:

* Prior treatment with a MEK inhibitor
* Active infection requiring intravenous antibiotics
* Pregnant, lactating or breast feeding women
* Prior radiation therapy within the last 14 days
* Unwillingness or inability to comply with study and follow-up procedures.
* Any foods/supplements that are strong inhibitors or inducers of CYP3A are prohibited at least 7 days prior to initiation of and during study treatment
* History of or evidence of retinal pathology on ophthalmologic examination that is considered a risk factor for neurosensory retinal detachment, RVO, or neovascular macular degeneration
* The risk factors for RVO are listed below. Exclusion should be considered by clinical discretion if they have the following conditions:

  * Uncontrolled glaucoma with intra-ocular pressures > 21mmHg
  * Serum cholesterol ≥ Grade 2
  * Hypertriglyceridemia ≥ Grade 2
  * Hyperglycemia ≥ Grade 2
* History of clinically significant cardiac dysfunction, unless deemed to be the direct result of disease, including the following:

  * Current unstable angina
  * Symptomatic congestive heart failure of NYHA class 2 or higher
  * Uncontrolled hypertension ≥ Grade 2 (patients with a history hypertension controlled with anti-hypertensives to ≤ Grade 2 are eligible).
  * Left ventricular ejection fraction (LVEF) below institutional lower limit of normal or below 50%
  * Uncontrolled arrhythmias
  * Myocardial infarction, severe/unstable angina, symptomatic congestive heart failure, cerebrovascular accident or transient ischemic attack within the previous 6 months

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2022-12-16 (Actual); Study Completion 2022-12-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eli Diamond, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (2):
- United States (2):
  - Mayo Clinic, Rochester, Minnesota
  - Memorial Sloan Kettering Cancer Center, New York, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Cobimetinib: This is an open-label, multicenter, phase II study exploring the efficacy and safety of single-agent Cobimetinib in patients with histiocytic disorders
Period: Overall Study
Arm/Group | Cobimetinib
Started | 35
Completed | 34
Not Completed | 1
Not completed — Not treated | 1

BASELINE CHARACTERISTICS:
Arm/Group | Cobimetinib
Number analyzed (Participants) | 35
Age, Continuous [Median (Full Range); unit: years] | 51 [18 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 34
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 27
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 35

OUTCOME MEASURES:

1. Primary Outcome: Best Overall Response
Description: by PET Response Criterial (PRC), with a dichotomous BOR of CR or PR versus neither of those. Assuming we use this binary endpoint of response, defined as best overall response of CR or PR versus not using the PET Response Criteria (PRC), a sample size of 18 patients provides 90% power to test the hypothesis that the response rate is promising (defined as 35% or higher) against a non-promising rate of 10% or lower.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Cobimetinib
Number analyzed (Participants) | 35
Participants
  Complete Metabolic Response | 21
  Partial Metabolic Response | 5
  Stable Metabolic Disease | 3
  Not evaluable | 6

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Cobimetinib
All-Cause Mortality (participants affected / at risk) | 8/35
Serious Adverse Events (participants affected / at risk) | 10/35
Other Adverse Events (participants affected / at risk) | 35/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cobimetinib (N=35)
Acute kidney injury (Renal and urinary disorders) | 4
Anemia (Blood and lymphatic system disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2
Cognitive disturbance (Nervous system disorders) | 2
Confusion (Psychiatric disorders) | 2
Constipation (Gastrointestinal disorders) | 2
Diarrhea (Gastrointestinal disorders) | 1
Fall (Injury, poisoning and procedural complications) | 1
Hypernatremia (Metabolism and nutrition disorders) | 4
Hyponatremia (Metabolism and nutrition disorders) | 2
Hypotension (Vascular disorders) | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3
Immune system disorders - Other (Immune system disorders) | 1
Infections and infestations - Other (Infections and infestations) | 2
Lung infection (Infections and infestations) | 2
Myocardial infarction (Cardiac disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Paroxysmal atrial tachycardia (Cardiac disorders) | 1
Platelet Count Decreased (Investigations) | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3
Retinal vascular disorder (Eye disorders) | 1
Sepsis (Infections and infestations) | 2
Spinal fracture (Injury, poisoning and procedural complications) | 2
Supraventricular tachycardia (Cardiac disorders) | 1
Syncope (Nervous system disorders) | 1
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Urinary tract infection (Infections and infestations) | 3
Vomiting (Gastrointestinal disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cobimetinib (N=35)
CPK Increased (Investigations) | 22
Rash acneiform (Skin and subcutaneous tissue disorders) | 22
Diarrhea (Gastrointestinal disorders) | 20
Anemia (Blood and lymphatic system disorders) | 19
Alanine aminotransferase increased (Investigations) | 16
Aspartate aminotransferase increasd (Investigations) | 16
Fatigue (General disorders) | 15
Hypomagnesemia (Metabolism and nutrition disorders) | 15
Lymphocyte count decreased (Investigations) | 15
Alkaline phosphatase increaseed (Investigations) | 14
Edema limbs (General disorders) | 13
Nausea (Gastrointestinal disorders) | 13
Pruritus (Skin and subcutaneous tissue disorders) | 13
White blood cell decreased (Investigations) | 12
Hypocalcemia (Metabolism and nutrition disorders) | 11
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 11
Hypoalbuminemia (Metabolism and nutrition disorders) | 10
Platelet count decreased (Investigations) | 10
Dry skin (Skin and subcutaneous tissue disorders) | 9
Hyponatremia (Metabolism and nutrition disorders) | 9
Blood bilirubin increased (Investigations) | 8
Constipation (Gastrointestinal disorders) | 8
Vomiting (Gastrointestinal disorders) | 8
Hypernatremia (Metabolism and nutrition disorders) | 7
Hypokalemia (Metabolism and nutrition disorders) | 7
Lipase increased (Investigations) | 7
Neutrophil count decreased (Investigations) | 7
Serum amylase increased (Investigations) | 7
Creatinine increased (Investigations) | 6
Dry mouth (Gastrointestinal disorders) | 6
Urinary tract infection (Infections and infestations) | 6
Activated partial thromboplastin time prolonges (Investigations) | 5
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5
Ejection fraction decreased (Cardiac disorders) | 5
Headache (Nervous system disorders) | 5
Hyperkalemia (Metabolism and nutrition disorders) | 5
Blurred vision (Eye disorders) | 4
Dyspepsia (Gastrointestinal disorders) | 4
Hypertension (Vascular disorders) | 4
Acute kidney injury (Renal and urinary disorders) | 3
Anorexia (Metabolism and nutrition disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Hyperglycemia (Metabolism and nutrition disorders) | 3
Hypoglycemia (Metabolism and nutrition disorders) | 3
Hypophosphatemia (Metabolism and nutrition disorders) | 3
Mucosal infection (Infections and infestations) | 3
Mucositis oral (Gastrointestinal disorders) | 3
Periorbital edema (Eye disorders) | 3
Alopecia (Skin and subcutaneous tissue disorders) | 2
Bloating (Gastrointestinal disorders) | 2
Bronchial infection (Infections and infestations) | 2
Conjunctivitis infective (Infections and infestations) | 2
Dizziness (Nervous system disorders) | 2
Edema face (General disorders) | 2
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2
Genital edema (Reproductive system and breast disorders) | 2
Hypotension (Vascular disorders) | 2
INR Increased (Investigations) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Oral pain (Gastrointestinal disorders) | 2
Pain (General disorders) | 2
Peripheral sensory neuropathy (Nervous system disorders) | 2
Purpura (Skin and subcutaneous tissue disorders) | 2
Skin infection (Infections and infestations) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-03): https://cdn.clinicaltrials.gov/large-docs/72/NCT02649972/Prot_SAP_000.pdf